CLINICAL TRIAL: NCT00690430
Title: A Multicenter, Randomized, Blinded Efficacy and Safety Study of Pasireotide LAR vs Octreotide LAR in Patients With Metastatic Carcinoid Tumors Whose Disease-related Symptoms Are Inadequately Controlled by Somatostatin Analogues.
Brief Title: Efficacy and Safety of Pasireotide Long Acting Release vs. Octreotide Long Acting Release in Patients With Metastatic Carcinoid Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CSOM230C2303; 2007-000739-25 (EudraCT Number)
Record Dates: First submitted 2008-05-15; First posted 2008-06-04 (Estimated); Results first posted 2013-07-30 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2013-06

CONDITIONS: Symptomatic Refractory Resistant Carcinoid Disease
Keywords: Carcinoid; neuroendocrine; gastroenteropancreatic; somatostatin analogue; Symptomatic Refractory Resistant Carcinoid Disease
MeSH Terms: conditions — Carcinoid Tumor | interventions — pasireotide; Octreotide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pasireotide LAR (Active Comparator): Patients assigned to pasireotide LAR will receive a 60 mg dose of pasireotide LAR i.m. depot injection once every 28 days (+/- 3 days) for 6 months at visits 2, 4, 5, 6, 7 and 8. A dose reduction to 40 mg is permitted if tolerability issues arise. In addition, after 24 hours of the first LAR injections the patients were permitted to use pasireotide s.c. formulation for breakthrough symptoms as needed.
  Interventions: Drug: Pasireotide
- Octreotide LAR (Active Comparator): Patients assigned to octreotide LAR will receive a 40mg dose of octreotide LAR i.m. depot injection once every 28 days (+/- 3 days) for 6 months at visits 2, 4, 5, 6, 7 and 8. A dose reduction to 30 mg is permitted if tolerability issues arise. Patients requiring a dose reduction are to return to the higher dose once the tolerability issue is resolved, if required for efficacy In addition, after 24 hours of the first LAR injections the patients were permitted to use octreotide s.c. formulation for breakthrough symptoms as needed.
  Interventions: Drug: Octreotide

INTERVENTIONS:
Drug: Pasireotide — Pasireotide LAR 60mg i.m. injection - patients may also receive pasireotide 600 µg s.c 3 times a day for symptom control as needed
  Other Names: SOM230
  Arms: Pasireotide LAR
Drug: Octreotide — Octreotide LAR 40mg i.m. depot injection - Patients may also receive octreotide 100 µg s.c. 3 times a day for symptom control as needed
  Other Names: Sadostatin LAR
  Arms: Octreotide LAR

SUMMARY:
The purpose of this randomized, multicenter, Phase III study was to compare the efficacy of paseriotide LAR and octreotide LAR in patients whose disease-related symptoms are inadequately controlled by currently available somatostatin analogues.

ELIGIBILITY:
Inclusion criteria:

* Male or female patients aged 18 or greater
* Patients with carcinoid tumors and symptoms (diarrhea and flushing) that are not adequately controlled by somatostatin analogues.
* Female patients of child bearing potential must have a negative pregnancy test at baseline.
* Patients for whom written informed consent to participate in the study has been obtained.

Exclusion criteria:

* Patients receiving radiolabeled somatostatin analogue therapy within the 3 months or any cytotoxic chemotherapy or interferon therapy within the 4 weeks prior to randomization
* Diabetic patients on anti-diabetic medications whose fasting blood glucose is poorly controlled as indicated by HBA1C > 8%
* Patients with symptomatic cholelithiasis
* Patient with malabsorption syndrome, short bowel or cholegenic diarrhea not controlled by specific therapeutic means.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2008-04; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (58):
- United States (10):
  - Scottsdale Healthcare/TGen Clinical Research Service TGen Clinical Research Service, Scottsdale, Arizona
  - University of Arizona / Arizona Cancer Center, Tucson, Arizona
  - Loma Linda University Dept. of Loma Linda CancerCent, Loma Linda, California
  - Cedars Sinai Medical Center Cedars Sinai 4, Los Angeles, California
  - H. Lee Moffitt Cancer Center/University of South Florida Dept of H. Lee Moffit, Tampa, Florida
  - Mount Sinai School of Medicine Study Coordinator, New York, New York
  - Montefiore Medical Center MMC, The Bronx, New York
  - Duke University Medical Center Dept. of Duke Cancer Center(2), Durham, North Carolina
  - St. Luke's Hospital and Health Network St. Luke's Cancer Network, Bethlehem, Pennsylvania
  - MD Anderson Cancer Center/University of Texas Dept. of MD Anderson (9), Houston, Texas
- Novartis Investigative Site, Buenos Aires, Buenos Aires, Argentina
- Austria (3):
  - Novartis Investigative Site, Graz
  - Novartis Investigative Site, Salzburg
  - Novartis Investigative Site, Vienna
- Belgium (2):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Ghent
- Novartis Investigative Site, Fortaleza, Ceará, Brazil
- Canada (3):
  - Novartis Investigative Site, Calgary, Alberta
  - Novartis Investigative Site, Halifax, Nova Scotia
  - Novartis Investigative Site, Montreal, Quebec
- France (7):
  - Novartis Investigative Site, Nice, France
  - Novartis Investigative Site, Strasbourg, France
  - Novartis Investigative Site, Clichy
  - Novartis Investigative Site, Dijon
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Montpellier
- Germany (6):
  - Novartis Investigative Site, Berlin, Germany
  - Novartis Investigative Site, Mainz, Germany
  - Novartis Investigative Site, Bad Berka
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, München
- Novartis Investigative Site, Jerusalem, Israel
- Italy (6):
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Modena, MO
  - Novartis Investigative Site, Perugia, PG
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Orbassano, TO
- Norway (2):
  - Novartis Investigative Site, Tromsø
  - Novartis Investigative Site, Trondheim
- Poland (2):
  - Novartis Investigative Site, Gdansk, Poland
  - Novartis Investigative Site, Gliwice, Silesian Voivodeship
- Novartis Investigative Site, Singapore, Singapore, Singapore
- Spain (2):
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Catalonia
  - Novartis Investigative Site, Santiago de Compostela, Galicia
- Sweden (5):
  - Novartis Investigative Site, Jönköping
  - Novartis Investigative Site, Linköping
  - Novartis Investigative Site, Lund
  - Novartis Investigative Site, Stockholm
  - Novartis Investigative Site, Uppsala
- United Kingdom (6):
  - Novartis Investigative Site, Withington, Greater Manchester
  - Novartis Investigative Site, Sheffield, South Yorkshire
  - Novartis Investigative Site, Basingstoke
  - Novartis Investigative Site, Birmingham
  - Novartis Investigative Site, Glasgow
  - Novartis Investigative Site, London

REFERENCES:
- See also: Visit NovartisClinicalTrials.com: Pre-qualify for a trial, and view a list of trials and participating study centers. — http://www.novartisclinicaltrials.com/etrials/searchTrial.do?trialID=679

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 186 patients were screened and 110 were randomized into the study.
Groups:
- Octreotide LAR: Patients assigned to octreotide LAR will receive a 40mg dose of octreotide LAR i.m. depot injection once every 28 days (+/- 3 days) for 6 months at visits 2, 4, 5, 6, 7 and 8. A dose reduction to 30 mg is permitted if tolerability issues arise. Patients requiring a dose reduction are to return to the higher dose once the tolerability issue is resolved, if required for efficacy. In addition, after 24 hours of the first LAR injections the patients were permitted to use octreotide s.c. formulation for breakthrough symptoms as needed.
- Extension: Octreotide LAR/Pasireotide LAR: After 6 month double blind core period, non-responders on Octreotide were given option to cross over to Pasireotide LAR in the Extension Phase of study.
Period: Core Phase
Arm/Group | Pasireotide LAR | Octreotide LAR | Extension: Octreotide LAR/Pasireotide LAR
Started | 53 ("Started" indicates Full Analysis Set (FAS) and Safety Set.) | 57 | 0 (This arm belongs to Extension Phase.)
Completed | 35 | 34 | 0
Not Completed | 18 | 23 | 0
Not completed — Abnormal Laboratory value | 0 | 1 | 0
Not completed — Adverse Event | 5 | 1 | 0
Not completed — Death | 0 | 2 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 3 | 0
Not completed — Subject no longer requires study drug | 1 | 0 | 0
Not completed — Lack of Efficacy | 8 | 10 | 0
Not completed — Administrative Problems | 0 | 1 | 0
Not completed — Early Termination | 0 | 5 | 0
Period: Extension Phase
Arm/Group | Pasireotide LAR | Octreotide LAR | Extension: Octreotide LAR/Pasireotide LAR
Started | 20 (Only those patients (except from UK) who received clinical benefit could extend therapy in extension) | 6 (Only those patients (except from UK) who received clinical benefit could extend therapy in extension) | 15 (Only those patients (except from UK) who received clinical benefit could extend therapy in extension)
Completed | 2 | 1 | 2
Not Completed | 18 | 5 | 13
Not completed — Lack of Efficacy | 3 | 1 | 4
Not completed — Abnormal Lab Values | 1 | 0 | 0
Not completed — Abnormal test procedure results | 1 | 0 | 0
Not completed — Administrative Problems | 0 | 1 | 1
Not completed — Adverse Event | 2 | 1 | 2
Not completed — Death | 1 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 2
Not completed — Early Termination | 10 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pasireotide LAR | Octreotide LAR | Total
Number analyzed (Participants) | 53 | 57 | 110
Age Continuous [Mean (Standard Deviation); unit: Years] | 61.2 (9.21) | 62.8 (11.91) | 62 (10.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 23 | 47
  Male | 29 | 34 | 63

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Who Achieved Clinical Symptom Improvement by Randomization Stratum and Treatment.
Description: Percentage of patients who received clinical benefit in symptom (diarrhea and/or flushing) improvement as: Diarrhea (D)+Flushing (F): Patients with a daily mean number (#) of at least four bowel movements and a total of five or more flushing episodes. Clinical Benefit Response Criteria (CBRC): <4 daily mean bowel movements AND at least 20% reduction from Baseline in the daily mean # of bowel movements AND any reduction in the total # of flushing episodes compared with Baseline. (D) Patients with a daily mean # of at least four bowel movements and a total # of <5 flushing episodes. (CBRC) <4 daily mean bowel movements AND at least a 20% reduction from Baseline in the daily mean # of bowel movements. (F) Patients with a total # of at least 14 flushing episodes and a daily mean # of <4 bowel movements (CBRC) At least a 30% reduction from Baseline in the total # of flushing episodes.
Time Frame: Month 6
Population: The Efficacy analyzable set consists of subset of FAS patients who were randomized at least six months prior to futility interim analysis data cut-off. It is for the primary efficacy analysis and secondary efficacy analysis except for tumor response assessment. Data reported was based on randomized patients at the time of the interim analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pasireotide LAR | Octreotide LAR
Number analyzed (Participants) | 43 | 45
Percentage of Participants
  Diarrhea and Flushing (N=37, 39) | 13.5 [4.5 to 28.8] | 28.2 [15.0 to 44.9]
  Diarrhea (N=2, 5) | 100 [15.8 to 100] | 20.0 [0.5 to 71.6]
  Flushing (N=4, 1) | 50 [6.8 to 93.2] | 0.0 [0.0 to 97.5]
  Overall (N=43, 45) | 20.9 [10.0 to 36.0] | 26.7 [14.6 to 41.9]

2. Secondary Outcome: Improvement in Daily Mean Number of Diarrhea Bowel Movement Episodes by Randomization Stratum and Treatment.
Description: Percent change from Baseline in mean daily bowel movements at Month 6 were compared between the two treatment groups using ANCOVA model with treatment as the main effect and symptom levels at Baseline (e.g. mean daily bowel movement at Baseline) and randomization stratum (D+F or D) as covariates. Percentage change = (Month 6 - baseline)/baseline.
Time Frame: 6 months
Population: The Efficacy analyzable set consists of the subset of FAS patients who were randomized at least six months prior to the futility DMC data cut-off. Patients who had symptoms at baseline and at 6 months were included in this analysis.
Measure: Mean (Standard Deviation); unit: Percentage of Episodes
Arm/Group | Pasireotide LAR | Octreotide LAR
Number analyzed (Participants) | 26 | 32
Percentage of Episodes
  Diarrhea and Flushing (N=24, 28) | -23.5 (24.28) | -38.4 (28.74)
  Predominantly Diarrhea (D) (N=2, 4) | -44.2 (10.26) | -22.9 (31.68)
  Overall (N=26, 32) | -25.1 (24.04) | -36.5 (29.05)

3. Secondary Outcome: Improvement in Daily Mean Number of Flushing Episodes by Randomization Stratum and Treatment.
Description: Percent change from Baseline in total number of flushing episodes comprising Month 6 were compared between the two treatment groups using ANCOVA model with treatment as the main effect and symptom levels at Baseline (e.g. total number of flushing episodes at Baseline) and randomization stratum (D+F or F) as covariates.
Time Frame: 6 months
Population: The Efficacy analyzable set consists of the subset of FAS patients who were randomized at least six months prior to the futility DMC data cut-off. Patients were analyzed according the treatment they were assigned to at randomization. (ITT) principle.
Measure: Mean (Standard Deviation); unit: Percentage of Episodes
Arm/Group | Pasireotide LAR | Octreotide LAR
Number analyzed (Participants) | 28 | 29
Percentage of Episodes
  Diarrhea and Flushing (N=24, 28) | -41.0 (41.06) | -52.8 (32.18)
  Predominately Flushing (N=4, 1) | -48.4 (23.13) | 47.2 (NA) — Standard Deviation could not be calculated because there was only 1 patient analyzed.
  Overall (N=28, 29) | -42.1 (38.76) | -49.4 (36.65)

4. Secondary Outcome: Pasireotide LAR vs. Octreotide LAR on Time to Symptom Response.
Time Frame: Month 6
Population: This Outcome Measure was planned in the protocol but not included in the analysis due to early termination of study due to lack of efficacy in symptom control.
Arm/Group | Pasireotide LAR | Octreotide LAR
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Objective Tumor Response Rate Assessed by Investigator
Description: Baseline evaluations were to include Triphasic CT scan or MRI of the abdomen. Triphasic CT or MRIs were to be read by same radiologist at each assessment, measuring the same target and non-target lesions and accounting for all lesions that were present at Baseline. All known disease was accounted for when assessing objective tumor status. Current objective tumor status was to be captured on Tumor Assessment CRF. Objective response rate was defined by RECIST criteria: Partial response (PR) must have ≥ 30% decrease in the sum of longest diameter of all target lesions, from the baseline sum. Complete response (CR) must have disappearance of all target and non-target lesions. For CR or PR, tumor measurements must be confirmed by 2nd assessments within 4 weeks. Progression = 20% increase in the sum of longest diameter of all target lesions, from smallest sum of longest diameter of all target lesions recorded at or after baseline; or a new lesion; or progression of non-target lesions.
Time Frame: Month 6
Population: Full Analysis Set (FAS) consists of all patients randomized into the study. Patients were analyzed according to the treatment they were assigned to at randomization. Patients randomized 6 months before the final clinical cutoff date were included in this analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pasireotide LAR | Octreotide LAR
Number analyzed (Participants) | 51 | 52
Percentage of Participants | 2.0 [0.0 to 10.4] | 3.8 [0.5 to 13.2]

6. Secondary Outcome: Pasireotide LAR vs. Octreotide LAR on Disease Control Rate Based on RECIST Criteria
Description: Disease control rate (DCR) is the proportion of patients with a best overall response of Complete Response (CR) or Partial Response (PR) or Stable Disease (SD). Complete Response (CR): Disappearance of all target lesions Partial Response (PR): At least a 30% decrease in the sum of the longest diameter of all target lesions, taking as reference the baseline sum of the longest diameters. Progressive Disease (PD): At least a 20% increase in the sum of the longest diameter of all measured target lesions, taking as reference the smallest sum of longest diameter of all target lesions recorded at or after baseline, or a new lesion; or progression of non-target lesions. Stable Disease (SD): Neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for PD. Unknown (UNK) Progression has not been documented and one or more target lesions have not been assessed or have been assessed using a different method than baseline.
Time Frame: Month 6
Population: Full Analysis Set (FAS) consists of all patients randomized into the study. Following the intent-to-treat principle, patients were analyzed according to the treatment they were assigned to at randomization. Patients with analyzable data at month 6 were included in this analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pasireotide LAR | Octreotide LAR
Number analyzed (Participants) | 51 | 52
Percentage of participants | 62.7 [48.1 to 75.9] | 46.2 [32.2 to 60.5]

7. Secondary Outcome: Pasireotide LAR vs. Octreotide LAR on Quality of Life Assessed by FACIT-D Questionnaire
Time Frame: Month 6
Population: as for outcome 4
Arm/Group | Pasireotide LAR | Octreotide LAR
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Pasireotide LAR vs. Octreotide LAR on Time to Symptom Progression
Time Frame: Month 6
Population: as for outcome 4
Arm/Group | Pasireotide LAR | Octreotide LAR
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Pasireotide LAR vs. Octreotide LAR on Duration of Symptom Response
Time Frame: Month 6
Population: as for outcome 4
Arm/Group | Pasireotide LAR | Octreotide LAR
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Assess the Proportion of Patients Who Achieved at Least a 30% Reduction in Frequency of Bowel Movements
Time Frame: Month 6
Population: as for outcome 4
Arm/Group | Pasireotide LAR | Octreotide LAR
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Groups:
- Extension Phase Pasireotide LAR: Patients assigned to pasireotide LAR will receive a 60 mg dose of pasireotide LAR i.m. depot injection once every 28 days (+/- 3 days) for 6 months at visits 2, 4, 5, 6, 7 and 8. A dose reduction to 40 mg is permitted if tolerability issues arise. In addition, after 24 hours of the first LAR injections the patients were permitted to use pasireotide s.c. formulation for breakthrough symptoms as needed.
- Extension Phase Octreotide LAR: Patients assigned to octreotide LAR will receive a 40mg dose of octreotide LAR i.m. depot injection once every 28 days (+/- 3 days) for 6 months at visits 2, 4, 5, 6, 7 and 8. A dose reduction to 30 mg is permitted if tolerability issues arise. Patients requiring a dose reduction are to return to the higher dose once the tolerability issue is resolved, if required for efficacy In addition, after 24 hours of the first LAR injections the patients were permitted to use octreotide s.c. formulation for breakthrough symptoms as needed.
- Crossover to Pasireotide LAR: After 6 month double blind core period, non-responders on Octreotide were given option to cross over to Pasireotide LAR in the Extension Phase of study.
Arm/Group | Pasireotide LAR | Octreotide LAR | Extension Phase Pasireotide LAR | Extension Phase Octreotide LAR | Crossover to Pasireotide LAR
Serious Adverse Events (participants affected / at risk) | 15/53 | 19/57 | 9/20 | 2/6 | 7/15
Other Adverse Events (participants affected / at risk) | 50/53 | 48/57 | 19/20 | 5/6 | 12/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pasireotide LAR (N=53) | Octreotide LAR (N=57) | Extension Phase Pasireotide LAR (N=20) | Extension Phase Octreotide LAR (N=6) | Crossover to Pasireotide LAR (N=15)
Carcinoid heart disease (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Endocardial fibrosis (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Tricuspid valve incompetence (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 3 | 1 | 0 | 1
Anorectal disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 4 | 1 | 1 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Intestinal infarction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Mesenteric vein thrombosis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 3 | 0 | 0 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Pneumoperitoneum (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 3 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 2 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0 | 0
Condition aggravated (General disorders) | 1 | 0 | 0 | 0 | 0
Device dislocation (General disorders) | 0 | 1 | 0 | 0 | 0
Device infusion issue (General disorders) | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 2 | 2 | 0 | 0 | 1
General physical health deterioration (General disorders) | 1 | 1 | 1 | 0 | 0
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 1 | 0 | 0 | 0
Medical device complication (General disorders) | 0 | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 2 | 0 | 1 | 0
Hepatomegaly (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 1
Clostridial infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Infectious peritonitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood bicarbonate decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 1 | 0 | 0 | 0
Blood pH increased (Investigations) | 1 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 1 | 1 | 0 | 0
Liver function test abnormal (Investigations) | 1 | 0 | 0 | 0 | 0
Troponin increased (Investigations) | 0 | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 2 | 2 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 2 | 1 | 1 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 0 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Carcinoid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Carcinoid tumour of the gastrointestinal tract (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Metastases to chest wall (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Metastatic carcinoid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Central nervous system lesion (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Nephritis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1
Renal failure chronic (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Urinary tract disorder (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Respite care (Social circumstances) | 0 | 0 | 1 | 0 | 0
Flushing (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Vein disorder (Vascular disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pasireotide LAR (N=53) | Octreotide LAR (N=57) | Extension Phase Pasireotide LAR (N=20) | Extension Phase Octreotide LAR (N=6) | Crossover to Pasireotide LAR (N=15)
Anaemia (Blood and lymphatic system disorders) | 3 | 1 | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Aortic valve sclerosis (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 3 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 2 | 1 | 0 | 0 | 1
Bundle branch block right (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Dilatation ventricular (Cardiac disorders) | 1 | 0 | 1 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 1 | 1 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 5 | 0 | 0 | 2
Pulmonary valve incompetence (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Tricuspid valve incompetence (Cardiac disorders) | 2 | 3 | 1 | 0 | 2
Birth mark (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 0 | 2 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 1 | 0 | 0
Dry eye (Eye disorders) | 2 | 0 | 1 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 1 | 0 | 0
Glaucoma (Eye disorders) | 0 | 0 | 0 | 0 | 1
Visual impairment (Eye disorders) | 0 | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 3 | 1 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 8 | 8 | 1 | 0 | 3
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 3 | 2 | 1 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Anal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 4 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 12 | 9 | 4 | 0 | 2
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 3 | 3 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Faecal incontinence (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 7 | 1 | 2 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 3 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 2 | 4 | 0 | 0
Nausea (Gastrointestinal disorders) | 10 | 7 | 4 | 0 | 3
Painful defaecation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Proctalgia (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 2
Proctitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Rectal ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Short-bowel syndrome (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Varices oesophageal (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 7 | 4 | 0 | 3
Asthenia (General disorders) | 5 | 6 | 4 | 1 | 1
Chest pain (General disorders) | 1 | 1 | 0 | 0 | 2
Chills (General disorders) | 0 | 1 | 2 | 0 | 0
Fatigue (General disorders) | 11 | 8 | 6 | 1 | 3
General physical health deterioration (General disorders) | 0 | 0 | 1 | 0 | 0
Injection site pain (General disorders) | 0 | 1 | 0 | 0 | 1
Localised oedema (General disorders) | 0 | 0 | 1 | 0 | 0
Malaise (General disorders) | 0 | 4 | 0 | 0 | 0
Oedema peripheral (General disorders) | 9 | 5 | 5 | 0 | 3
Pain (General disorders) | 1 | 1 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 2 | 4 | 1 | 2
Biliary dilatation (Hepatobiliary disorders) | 1 | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 4 | 4 | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1 | 0
Biliary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 2 | 1 | 1 | 1 | 1
Candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 2 | 0 | 0 | 1
Gastrointestinal bacterial infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Incision site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 2 | 5 | 0 | 1 | 1
Sinusitis (Infections and infestations) | 1 | 1 | 1 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 3 | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 2 | 0 | 1 | 2
Viral infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 3 | 1 | 0 | 1
Albumin urine present (Investigations) | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 3 | 2 | 0 | 2
Bilirubin conjugated increased (Investigations) | 0 | 1 | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 2 | 5 | 2 | 0 | 2
Blood bilirubin increased (Investigations) | 2 | 0 | 1 | 0 | 0
Blood calcium increased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 3 | 3 | 2 | 0 | 1
Blood glucose increased (Investigations) | 3 | 0 | 1 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood magnesium decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood testosterone decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood triglycerides increased (Investigations) | 1 | 0 | 0 | 0 | 2
Blood urea increased (Investigations) | 0 | 1 | 1 | 0 | 0
Blood urine present (Investigations) | 0 | 0 | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 3 | 2 | 0 | 2
Glycosylated haemoglobin increased (Investigations) | 0 | 0 | 0 | 0 | 1
Haematocrit increased (Investigations) | 0 | 1 | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 1 | 1 | 0 | 0 | 1
Haemoglobin increased (Investigations) | 0 | 0 | 0 | 0 | 1
Red blood cell count increased (Investigations) | 0 | 1 | 0 | 0 | 1
Weight decreased (Investigations) | 8 | 4 | 2 | 0 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 4 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 2 | 2 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 6 | 0 | 0 | 0 | 0
Glucose tolerance impaired (Metabolism and nutrition disorders) | 2 | 1 | 2 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 15 | 3 | 7 | 1 | 2
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 1 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 3 | 3 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 3 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Increased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 3 | 1 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 3 | 3 | 0 | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 | 1 | 2 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 4 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 0 | 1 | 0 | 2
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Aphonia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Cervicobrachial syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 5 | 1 | 4 | 0 | 0
Dysaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Headache (Nervous system disorders) | 7 | 1 | 2 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 1 | 0 | 0
Lethargy (Nervous system disorders) | 3 | 0 | 0 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Muscle contractions involuntary (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 2 | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 2 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 3 | 3 | 2 | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 3 | 1 | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 3 | 0 | 0 | 3
Libido decreased (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 2 | 0 | 1 | 0
Glycosuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 1 | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 2 | 1 | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 1 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 3 | 2 | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0 | 0
Reflux laryngitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 3 | 1 | 1 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 3 | 1 | 0 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 4 | 1 | 2 | 0 | 2
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Alcohol use (Social circumstances) | 0 | 0 | 1 | 0 | 0
Axillary vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Flushing (Vascular disorders) | 5 | 4 | 0 | 0 | 2
Hypertension (Vascular disorders) | 3 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 1 | 2 | 0 | 1
Lymphoedema (Vascular disorders) | 0 | 1 | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 1
Subclavian vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Thrombophlebitis superficial (Vascular disorders) | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators are NOT employed by the organization sponsoring the study. Other disclosure agreement that restricts the right of the PI to discuss or publish trial results after the trial is completed. The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial.